



## **Participant Informed Consent Form**

| RAS ID: | 320293 | | | |
|---|---|---|---|---|
| Trial Name: | Evaluation of Pilot Online Bi 18s. | nge Eating Diso | rder Group Intervention | for under |
| Chief<br>nvestigator:<br>Principal<br>nvestigator: | Dominique Muhumuza | | | |
| | Dominique Muhumuza | | | |
| Participant Ide | ntification | | | |
| number: | | | | |
| | | | | Please<br>initial |
| 1. I confirm th | nat I have: | | | each box |
| | nderstand the information sheet <b>PIS</b> for the above study. | Parent Carer -BE G | roup Intervention | |
| | n time to think whether or not I want r<br>swers that I think are reasonable. | myself and my child | to take part, ask questions | |
| have been | I that this study is designed to further<br>approved by the Research Ethics Co<br>Ethics Committee of Coventry and Wa | mmittee of Newmar | university and by the | |
| | nd that my taking part is voluntary and ing any reason, without my medical o | | | |
| | ry and complete the questionnaires. them if I wish. | I understand that I | can take a break or stop | |
| 4. I understar | nd that: | | | |
| My child wi | II be participating in a group intervent | tion | | |
| I will be ask | ked support my child to complete wee | ekly tasks as part of | the group | |
| • I will be ask | ked to attend an information session | | | |
| I understand that my questionnaires and feedback may be looked at by people from the Coventry and Warwickshire Partnership trust or Newman University. I give permission for these individuals to have access to all information collected. | | | | |
| 6. I understand that information collected will be kept confidential. However, if I tell the researchers something they think is likely to result in immediate harm to myself or others, they may have to talk to me about disclosing this in line with the law and local safeguarding procedures. | | | | |
| 7. I agree for | the ED team to inform my child's GP | that I am participati | ng in this project. | |
| 8. I agree to t | ake part in the above study. | | | |
| Your name (in o | capitals) | Date | Signature | |
| Name of person | n taking consent (in capitals) | Date | Signature | |
| Name of person | rtaking consent (iii capitals) | | Originature | |
| Nama | | Doto | Cinnatura | |
| (in capitals) | recording consent (if different) | Date | Signature | |

When completed, the original should be kept in the Investigator Site File, a copy should be given to the patient and one kept in the study notes along with the Participant Information Sheet.

ICF Parent/Carer - BE Group Intervention 2022.docx

Version 1: 08/02/2023 Page 1 of 1